CLINICAL TRIAL: NCT00863642
Title: Early Versus Delayed Surgery for Gallstone Pancreatitis: A Prospective Randomized
Brief Title: Early Versus Delayed Surgery for Gallstone Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, christian de virgilio, Professor of Surgery, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12935-01
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Gallstone Pancreatitis
Keywords: Early cholecystectomy; gallstone pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early (Experimental): In patients who present with mild to moderate gallstone pancreatitis, those randomized to the early arm will undergo laparoscopic cholecystectomy within 48 hours of admission, regardless of laboratory values normalization and resolution of abdominal pain.
  Interventions: Procedure: Laparoscopic cholecystectomy within 48 hours of admission
- Control (Other): In patients in the control arm, laparoscopic cholecystectomy is delayed until laboratory values normalize and abdominal pain resolves.
  Interventions: Procedure: Laparoscopic cholecystectomy after resolution of abdominal pain and laboratory values

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy within 48 hours of admission — Patients are taken to the operating room for laparoscopic cholecystectomy within 48 hours of admission
  Arms: Early
Procedure: Laparoscopic cholecystectomy after resolution of abdominal pain and laboratory values — Patients are taken to the operating room for laparoscopic cholecystectomy after resolution of abdominal pain and laboratory values
  Arms: Control

SUMMARY:
While there exists consensus among surgeons that patients with gallstone pancreatitis should undergo cholecystectomy to prevent recurrence, the precise timing of laparoscopic cholecystectomy for mild to moderate disease remains controversial. We hypothesize that laparoscopic cholecystectomy performed within 48 hours of admission, regardless of resolution of abdominal pain or abnormal laboratory values, will result in a shorter hospital stay.

DETAILED DESCRIPTION:
Acute pancreatitis is a common diagnosis worldwide, with more than 220,000 cases reported annually in the United States alone. The leading etiology is gallstones.1 Gallstone pancreatitis is thought to occur due to transient obstruction of the common channel that drains both the biliary and pancreatic ducts, resulting in inflammation of the pancreas. The pancreatitis that ensues is usually mild and self-limited and the treatment is initially supportive with subsequent laparoscopic cholecystectomy (LC). However, a small subgroup of patients develop severe pancreatitis and/or concomitant cholangitis. When the latter is present, ERC and sphincterotomy with stone extraction as indicated are typically performed.

While there is a clear consensus that patients who present with gallstone pancreatitis should undergo cholecystectomy to prevent recurrence, precise timing of surgery remains controversial. In patients with severe pancreatitis (Ranson's > 3), there is consensus that surgery is delayed until the pancreatitis has resolved because early operation is associated with a higher complication rate. 2 However, despite more than 30 years of debate in the surgical literature, the optimal timing of surgery in mild to moderate pancreatitis (Ranson's ≤ 3) remains unclear. With recurrence rates for gallstone pancreatitis reported as high as 63%3 and with some of the repeat attacks occurring within two weeks of initial index presentation1, most investigators have recommended cholecystectomy during the initial hospitalization.4,5 Still, the actual timing of surgery during the initial index hospitalization is unsettled. In practice, surgeons often delay surgery until there is evidence of complete resolution of the inflammatory process, as evidenced by absence of abdominal pain and normalization of liver functional tests and pancreatic enzymes.6 Unfortunately, this strategy may result in prolongation of hospitalization without any proven benefit.

A previous prospective, non-randomized study from our institution suggested that early cholecystectomy could safely be performed within 48 hours of admission in patients with mild to moderate pancreatitis, regardless of resolution of abdominal pain and abnormal laboratory values. In this study, when compared to a retrospective control group in which surgery was delayed until there was resolution of clinical and laboratory parameters, hospital stay was significantly reduced from a median of 7 days to 4 days, without additional complications.7 In order to address the optimal timing of surgery in a more definite fashion, a prospective randomized study was performed in which patients with mild to moderate gallstone pancreatitis were allocated to either an early group (surgery within 48 hours of presentation) or a control group (surgery after resolution of abdominal pain and normalization of laboratory values) and assessed overall outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All adults are included between the age of 18 and 100 with mild to moderate gallstone pancreatitis.
* A subject is classified as having gallstone pancreatitis if they had the following:

  1. upper abdominal pain, nausea, vomiting and epigastric tenderness;
  2. absence of ethanol abuse;
  3. elevated amylase level to at least twice the upper limit of normal and elevated lipase level to at lease three times the upper limit of normal; and
  4. imaging confirmation of gallstones.
* The classification of mild to moderate pancreatitis is defined by the presence of the following:

  1. three or fewer Ranson's criteria on admission: age > 55 years, glucose > 200 mg/dL , LDH> 350 mg/dL, AST > 250 units/L, and WBC>16 K/mm3;
  2. clinical stability with admission to a non-monitored ward bed;
  3. absence of acute cholangitis: defined as a temperature >38.6°C, right upper quadrant pain and tenderness, and significant hyperbilirubinemia; and
  4. low suspicion for a retained common bile duct (CBD) stone (total bilirubin <4 mg/dl on admission).

Exclusion Criteria:

* Severe pancreatitis (as defined by the presence of more than three Ranson's criteria on admission);
* Suspected concomitant acute cholangitis;
* High suspicion for retained common bile duct stone (total bilirubin ≥ 4 mg/dl on admission or ultrasound demonstration of CBD stone);
* Patient refusal to participate;
* Severe preexisting medical comorbidities contraindicating cholecystectomy (as determined by the primary physicians);
* Pregnancy,
* Prior gastric bypass surgery (making ERC difficult )
* Admission to a monitored unit. The need for admission to a monitored bed is determined by the admitting surgeon and is guided primarily by a need for aggressive fluid administration as demonstrated by severe volume depletion (e.g., admission tachycardia >110 beats/minute, blood urea nitrogen > 15 mg/dl) or evidence of cholangitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Days in the hospital

SECONDARY OUTCOMES:
Rates of conversion to open surgery, complication rates and rates of need for endoscopic retrograde cholangiogram | Within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Harbor-UCLA Medical Center, Torrance, California, United States

REFERENCES:
- [Background] Rosing DK, de Virgilio C, Yaghoubian A, Putnam BA, El Masry M, Kaji A, Stabile BE. Early cholecystectomy for mild to moderate gallstone pancreatitis shortens hospital stay. J Am Coll Surg. 2007 Dec;205(6):762-6. doi: 10.1016/j.jamcollsurg.2007.06.291. Epub 2007 Sep 17. PMID 18035259
- [Derived] Aboulian A, Chan T, Yaghoubian A, Kaji AH, Putnam B, Neville A, Stabile BE, de Virgilio C. Early cholecystectomy safely decreases hospital stay in patients with mild gallstone pancreatitis: a randomized prospective study. Ann Surg. 2010 Apr;251(4):615-9. doi: 10.1097/SLA.0b013e3181c38f1f. PMID 20101174